CLINICAL TRIAL: NCT02662608
Title: NOTCH 1 Inhibitor Brontictuzumab for Adenoid Cystic Carcinoma Bearing Two Activating NOTCH1 Mutations
Brief Title: Compassionate Use of Brontictuzumab for Adenoid Cystic Carcinoma (ACC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIND15-0074
Record Dates: First submitted 2016-01-22; First posted 2016-01-25 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Adenoid Cystic Carcinoma
Keywords: Brontictuzumab
MeSH Terms: conditions — Carcinoma, Adenoid Cystic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brontictuzumab (Experimental): 1.5 mg/Kg of Brontictuzumab single agent intravenously every three weeks.
  Interventions: Drug: Brontictuzumab

INTERVENTIONS:
Drug: Brontictuzumab — 1.5 mg/Kg intravenously every three weeks.
  Other Names: OMP-52M51

SUMMARY:
The goal of this study is to start treatment with the NOTCH1 inhibitor brontictuzumab in an attempt to control tumors and prolong survival. The therapy involves participant being given the drug brontictuzumab to treat adenoid cystic carcinoma (ACC) with NOTCH 1 mutations. This is considered an investigational treatment.

DETAILED DESCRIPTION:
Treatment:

Participant will receive brontictuzumab by vein over 30 minutes one time every 3 weeks.

Clinic Visits:

On Day 1 of Cycle 1 and then every 3 weeks from then on:

* Participant will have a physical exam
* Blood (about 3 teaspoons) will be drawn for routine tests.

Every 6 weeks, participant will have an MRI and CT scan to check the status of the disease.

Length of Treatment:

Participant may continue taking brontictuzumab for as long as the doctor thinks it is in their best interest. Participant will no longer be able to take the drug if the disease gets worse, they develop another illness that prevents receiving more treatment, or if intolerable side effects occur.

Brontictuzumab is not FDA approved or commercially available. It is currently being used for research purposes only.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
2. Organ and marrow function as follows: absolute neutrophil count (ANC) ≥1000/mm3, platelets ≥50,000/dL, hemoglobin ≥8 g/dL, bilirubin ≤ 1.5 times the upper limit of normal, serum creatinine ≤1.5 mg/dL or creatinine clearance ≥50 mL/min, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal.
3. Central Nervous System (CNS) metastases allowed if subject does not require steroids, brain metastases are clinically stable without symptomatic progression
4. Capability to understand and comply with the protocol and signed informed consent document.

Exclusion Criteria:

1. Major medical conditions that might affect study participation (e.g. uncontrolled pulmonary, renal, or hepatic dysfunction, uncontrolled infection, cardiac disease)
2. Inability or unwillingness to abide by the study protocol or cooperate fully with the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-12-29 (Actual); Primary Completion 2016-03-06 (Actual); Study Completion 2016-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renata Ferrarotto, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment was limited to single participant compassionate use in December 2015.
Groups:
- Brontictuzumab: Brontictuzumab 1.5 mg/Kg intravenously every 3 weeks.
Period: Overall Study
Arm/Group | Brontictuzumab
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Brontictuzumab
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disease Progression
Description: Tumor response for measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) to establish disease progression. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Brontictuzumab
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse event collection with three week treatment cycle.
Arm/Group | Brontictuzumab
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brontictuzumab (N=1)
Diarrhea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes